CLINICAL TRIAL: NCT02566083
Title: Post-Approval Study of the Tecnis® Toric IOL, Models ZCT300 and ZCT400
Brief Title: Post-Approval Study of the Tecnis® Toric IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIOL-202-TPAS
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- non-toric intraocular lens (Active Comparator): non-toric approved intraocular lens
  Interventions: Device: non-toric intraocular lens
- toric intraocular lens (Active Comparator): approved toric intraocular lens
  Interventions: Device: toric intraocular lens

INTERVENTIONS:
Device: non-toric intraocular lens — TECNIS One-piece Monofocal Model ZCB00
  Arms: non-toric intraocular lens
Device: toric intraocular lens — TECNIS One-piece Toric Models ZCT300 or ZCT400
  Arms: toric intraocular lens

SUMMARY:
This study is a prospective, multicenter, bilateral, non-randomized, open-label, comparative clinical study conducted at up to 80 sites in the USA. Subjects will choose to be bilaterally implanted with either 1) the TECNIS 1-Piece Toric IOLs, Model ZCT300 and/or ZCT400, or 2) the TECNIS Monofocal Model ZCB00 non-toric control IOL, according to subject preference

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age
* Bilateral cataracts
* Preoperative keratometric cylinder in both eyes
* Most appropriate toric IOL model choice (ZCT300 or ZCT400)
* Predicted residual refractive cylinder, based on the AMO Toric IOL Calculator, must be:

  ≤ 0.69 D for a ZCT300 IOL or ≤ 0.88 D for a ZCT400 IOL
* Clear intraocular media other than cataract in each eye
* Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visits
* Ability to understand, read and write English in order to consent to study participation and complete a study questionnaire
* Signed informed consent and HIPAA authorization

Exclusion Criteria:

* Irregular corneal astigmatism
* Any corneal pathology/abnormality other than regular corneal astigmatism
* Previous corneal surgery
* Recent ocular trauma or intraocular surgery that is not resolved/stable or may affect visual outcomes
* Any pupil abnormalities
* Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration, including pseudoexfoliation, trauma, or posterior capsule defects
* Known ocular disease or pathology that may affect visual acuity or that may require surgical intervention during the course of the study
* Concurrent participation or participation during 30 days prior to preoperative visit in any other clinical study
* Planned monovision correction
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2019-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devi Priya Janakiraman, OD, FAAO, Study Director — Johnson & Johnson Surgical Vision
Locations (44):
- United States (44):
  - Eye Center South, Dothan, Alabama
  - Arizona Eye Cente, Chandler, Arizona
  - Fishkind, Bakewell & Maltzman Eye Care & Surgery Cente, Tucson, Arizona
  - Boozman-Hof Regional Eye Clinic, Rogers, Arkansas
  - Empire Eye & Laser Center, Bakersfield, California
  - Atlantis Eye Care, Huntington Beach, California
  - Scripps Clinic Medical Group, La Jolla, California
  - Southern California Eye Physicians & Associates, Long Beach, California
  - Feinerman Vision Center, Newport Beach, California
  - Coastal Vision, Orange, California
  - California Eye Medical Specialists, Pasadena, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - Katzen Eye Care & Laser Center, Boynton Beach, Florida
  - The Eye Associates, Bradenton, Florida
  - Cape Coral Eye Center, Cape Coral, Florida
  - Levenson Eye Associates, Inc., Jacksonville, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Virdi Eye Clinic & Laser Vision Center, Rock Island, Illinois
  - Senior Health Services, Louisville, Kentucky
  - Chesapeake Eye Care and Laser Center, Annapolis, Maryland
  - Solomon Eye Associates, Bowie, Maryland
  - Eye Doctors of Washington, Chevy Chase, Maryland
  - Oakland Ophthalmic Surgery, P.C., Birmingham, Michigan
  - TLC Eye Care and Laser Centers, Chelsea, Michigan
  - Mercy Clinic Eye Specialist, Springfield, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Ophthalmology Consultants, St Louis, Missouri
  - Kindermann Eye Associates, Cherry Hill, New Jersey
  - Matossian Eye Associates, Pennington, New Jersey
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - Pamel Vision & Laser Group, New York, New York
  - Fine, Hoffman & Sims, Eugene, Oregon
  - The Eye Center of Central PA, Allenwood, Pennsylvania
  - Ludwick Eye Center, Chambersburg, Pennsylvania
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Carolina Cataract & Laser Center, Ladson, South Carolina
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Loden Vision Centers, Goodlettsville, Tennessee
  - Houston Eye Associates, Houston, Texas
  - Whitsett Vision Group, Houston, Texas
  - Focal Point Vision, San Antonio, Texas
  - San Antonio Eye Specialists, San Antonio, Texas
  - Clarus Eye Centre, Lacey, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Toric IOL: Experimental (ZCT300, ZCT400)
- Non-toric IOL: Control (ZCB00)
Period: Overall Study
Arm/Group | Toric IOL | Non-toric IOL
Started | 214 | 151
Completed | 198 | 141
Not Completed | 16 | 10

BASELINE CHARACTERISTICS:
Population: All subjects who have at least one eye implanted with the study IOL (Toric or control) are included in the demographic analysis. For questionnaire results only subjects who were bilaterally implanted with study IOL (Toric or control) were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Toric IOL | Non-toric IOL | Total
Number analyzed (Participants) | 214 | 151 | 365
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (9.6) | 69.7 (10.0) | 69.5 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 82 | 202
  Male | 94 | 69 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 10 | 29
  Not Hispanic or Latino | 195 | 141 | 336
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 18 | 28
  White | 197 | 128 | 325
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Severe Visual Distortions
Description: The rate of severe visual distortions under overall circumstances for the five visual distortion items of interest (lines that slant, tilt, split or separate; flat surfaces appearing curved; objects appearing further away or closer than they are; objects appearing to have a different size or shape; and physical discomfort related to vision). The six month data were used for this endpoint if available and if not an earlier visit was used. If a subject had a lens repositioning the questionnaire prior to the repositioning was used if available.
Time Frame: 6 months
Population: All subjects bilaterally implanted with a toric IOL (ZCT300 or ZCT400) and all subjects bilaterally implanted with a control IOL (ZCB00). All subjects who were monocularly implanted with a toric IOL (ZCT300/400) or control were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Toric IOL | Non-toric IOL
Number analyzed (Participants) | 189 | 144
Participants
  With No severe visual distortion | 189 | 142
  With severe visual distortion | 0 | 2

ADVERSE EVENTS:
Time Frame: All AEs were reported and followed until resolution with a timeframe of 6 months. Subjects who reported IOL repositioning or severe visual distortion on the 6 month visit were followed up until 1 year postoperative.
Arm/Group | Toric IOL | Non-toric IOL
All-Cause Mortality (participants affected / at risk) | 1/214 | 2/151
Serious Adverse Events (participants affected / at risk) | 32/214 | 16/151
Other Adverse Events (participants affected / at risk) | 0/214 | 1/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toric IOL (N=214) | Non-toric IOL (N=151)
Lens repositioning (Surgical and medical procedures) | 12 (12) | 0 (0)
Epiretinal membrane with significant Vitreo-Retinal traction (Eye disorders) | 1 (1) | 0 (0)
Cystoid Macular Edema (Eye disorders) | 6 (8) | 5 (5)
Macular Hole (Eye disorders) | 1 (1) | 0 (0)
Clinically Significant Macular Edema (Eye disorders) | 0 (0) | 1 (1)
Residual Cortical material (Surgical and medical procedures) | 1 (1) | 1 (1)
Elevated intraocular pressure requiring treatment (Eye disorders) | 2 (2) | 0 (0)
Capsular Rupture (Eye disorders) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0)
Hyphema (Eye disorders) | 1 (1) | 0 (0)
Macular Edema (Eye disorders) | 1 (1) | 0 (0)
Capsular Tear (Eye disorders) | 1 (1) | 0 (0)
Vitreous Strand (Eye disorders) | 1 (1) | 0 (0)
Hospitalization (General disorders) | 2 (2) | 8 (9)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Death (General disorders) | 1 (1) | 2 (2)
Crerebrovascular Accident (Vascular disorders) | 1 (1) | 0 (0)
Ulcerative Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toric IOL (N=214) | Non-toric IOL (N=151)
Cystoid Macular Edema (Eye disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at any time.

DOCUMENTS (2):
  • Study Protocol (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT02566083/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT02566083/SAP_001.pdf